CLINICAL TRIAL: NCT05298553
Title: Diagnostic Accuracy of WEARable TECHnology Single-lead ECG in Detecting Cardiac Arrhythmias: WEAR-TECH ECG
Brief Title: Diagnostic Accuracy of WEARable TECHnology Single-lead ECG in Detecting Cardiac Arrhythmias
Acronym: WEAR-TECH ECG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: University Hospital Birmingham (Other); University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Tim Betts MD MBChB FRCP, Primary Investigator, Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 15487
Record Dates: First submitted 2021-12-12; First posted 2022-03-28 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Cardiac Arrhythmia; Atrial Fibrillation
Keywords: Apple Watch;; Skylabs CART-I Ring; Wearable Devices
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): The order in which the wearable devices being investigated will be randomly assigned in a 1:1 fashion.
  Simultaneous 12-lead ECG and single-lead ECG with the SkyLabs CART-I ring followed by the Apple Watch.
  Interventions: Device: Group A
- Group 2 (Experimental): The order in which the wearable devices being investigated will be randomly assigned in a 1:1 fashion.
  Simultaneous 12-lead ECG and single-lead ECG with the Apple Watch followed by the SkyLabs CART-I ring.
  Interventions: Device: Group B

INTERVENTIONS:
Device: Group A — Participants will be asked to perform a simultaneous 30-seconds 12-lead ECG and single-lead ECG for each wearable device: Skylab CART-I ring followed by Apple Watch.
  Arms: Group 1
Device: Group B — they will be asked to perform a simultaneous 30-seconds 12-lead ECG and single-lead ECG for each wearable device: Apple Watch followed by the Skylab CART-I ring.
  Arms: Group 2

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia (irregular heart rhythm), affecting 1-2 million people in the UK. AF significantly increases the risk of an AF-related stroke, heart failure and dementia. A significant proportion of people will have no symptoms, and they may only be found to have AF after suffering an AF-related stroke.

An electrocardiogram (ECG) uses sensors placed on the skin to record the heart's electrical activity. A 12-lead ECG uses 10 sensors and is the gold-standard (best available test) to detect any abnormal heart rhythm disturbances. Until recently, a 12-lead ECG showing an irregular heart rhythm was required to make a diagnosis of AF but as AF episodes are often short and unpredictable it may be missed. Therefore, a small device that continuously records heartbeat and heart rhythm could make the diagnosis of arrhythmias and AF much quicker and easier.

Accessories such as watches or rings - referred to as wearable devices - have extremely good sensors that measure pulse rate by detecting small changes in skin colour during each heartbeat and can perform a single-lead ECG. Algorithms built in the wearable devices can identify irregular heart rhythms, such as atrial fibrillation.

The purpose of this study is to test two new wearable devices - the Skylabs CART-I ring and the Apple Watch - in detecting abnormal heart rhythm recording and recording ECGs. The investigators plan to recruit 500 patients attending Cardiology Departments in several hospitals in the UK and will ask them to wear the Apple Watch and the CART-I and perform 12-lead ECG with each device (two in total). No extra follow-up visits are required. At the end of the study, the investigators will compare interpretation by two cardiologists of the wearable devices' ECGs and the 12-lead ECGs and look at their ability to automatically detect abnormal rhythms.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Male or female aged 18 years or above.
* Indication for 12-lead ECG.

Exclusion Criteria:

* Unable to comply with instructions.
* Tattoos in the wrists or fingers where the device will be placed.
* Severe skin allergy to silicone (Apple Watch wrist band) or nickel allergies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Compare the accuracy of physician rhythm interpretation of 1-lead ECG generated by SkyLabs CART-I ring and Apple Watch versus 12-lead ECG (gold-standard) | 1 Day
  Assessment of diagnostic accuracy of SkyLabs CART-I ring and Apple Watch 1-lead ECGs interpretation for different cardiac arrhythmias (atrial compared with a 12-lead ECG (gold-standard).

SECONDARY OUTCOMES:
Compare the accuracy of automatic AF detection of the SkyLabs CART-I Ring and Apple Watch versus a cardiologist interpretation of a 12-lead ECG (gold-standard) | 1 Day
  Assessment of diagnostic accuracy of the AF detection algorithm of the Skylab CART-I ring and Apple Watch compared to a 12-lead ECG (gold-standard).
Compare the accuracy of ECG interval measurement for the SkyLabs CART-I Ring and Apple Watch to a 12-lead ECG (gold-standard) | 1 Day
  Level of agreement of measured interval duration between the SkyLabs CART-I ring, Apple Watch 1-lead ECG and a 12-lead ECG.
Compare the accuracy of heart rate detection of the SkyLabs CART-I ring and Apple Watch 1-lead ECG to a 30-second 12-lead ECG | 1 Day
  Correlation coefficient between the mean heart rate from simultaneous single lead and 12 lead ECG acquisitions.
Compare the accuracy of rhythm interpretation of SkyLabs CART-I ring 1-lead ECG to combined PPG (plethosysmography) signal and 1-lead ECG. | 1 Day
  Assessmen of diagnostic accuracy of the Skylab CART-I ring if a PPG signal is added.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Betts, MD, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (3):
- United Kingdom (3):
  - Oxford Univeristy Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - University Hospital Birmingham, Birmingham
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: Undecided